CLINICAL TRIAL: NCT06884046
Title: Evaluation of the Feasibility of Support for the Management of Parental Stress in Surgical Resuscitation of Congenital Heart Diseases
Brief Title: Support for the Management of Parental Stress in Surgical Resuscitation of Congenital Heart Diseases
Acronym: Et APRéS Ca
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2022/78; 2024-A00681-46 (Other: ID-RCB number)
Record Dates: First submitted 2025-02-25; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-02

CONDITIONS: Complex Congenital Heart Disease
Keywords: Neurodevelopment; Stress parental; Parental guidance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Accompaniment project (Experimental): The experimental intervention envisaged combines specific monitoring and the implementation of a personalised support programme.
  Interventions: Other: Personalized support project

INTERVENTIONS:
Other: Personalized support project — 1. Presence of a child nurse at the consultation of the anesthesiologist-resuscitator.
  2. Antenatal paramedical consultation conducted by a child nurse composed of a semi-structured interview and an evaluation of Parental Stress by the ISP-4 self-questionnaire.
  3. Implementation of the personalized support project
  4. Self-assessment of parental stress using the ISP-4 self-questionnaire (child admitted to intensive care or resuscitation unit)
  5. Application of the personalised support project
  6. Self-assessment of parental stress using the ISP-4 self-questionnaire (child discharged from intensive care)
  7. Paramedical follow-up consultation with parents (semi-directive interview, ISP-4 self-questionnaire) and assessment of the child's psychomotor development in the child's 6th month of life

SUMMARY:
Half of children with congenital heart disease develop specific neurodevelopmental disorders. Neurodevelopmental disorders are the leading cause of morbidity in these children. They can be increased by perioperative complications, the family and economic socio-economic environment and the level of parental stress. The stress perceived by parents of children with congenital heart disease varies depending on the time of diagnosis, the organization of care inherent in neonatal management and the type of pathology diagnosed.

The main objective is to evaluate the feasibility of a multidisciplinary and personalised model of support for parental stress, from the ante-natal period, in the context of their child's neonatal cardiac surgery.

DETAILED DESCRIPTION:
Congenital heart disease (CC) is the most common congenital malformation. Every year, 8 newborns out of 1000 are affected by these pathologies worldwide and about 20% of them will require intervention in the first days of life. The complexity of heart disease, factors intrinsic to the patient as well as surgical techniques can be the cause of neurological abnormalities. Indeed, 43% of these CC newborns are already carriers of a cerebral anomaly in the perinatal period.

Neurodevelopmental disorders (NDD) are the leading cause of morbidity in these children. They can be increased by perioperative complications, the family and economic socio-economic environment and the level of parental stress. The stress perceived by parents of children with CC varies depending on the time of diagnosis, the type of pathology and the organization of neonatal care.

It is essential to accompany these parents with personalized care. It must be comprehensive, multidisciplinary and empathetic, with the aim of improving the neurodevelopmental prognosis of these children, and family well-being.

Through this project of accompaniment proposed from the antenatal, we innovate by integrating consultations by the paramedical team of the resuscitation, the implementation of a personalized support project that meets the expectations and needs of families for better care of their child. A parental stress assessment will be carried out at 4 times of the family care journey.

ELIGIBILITY:
Inclusion Criteria:

* Parents whose fetus has congenital heart disease diagnosed in antenatal, which will be operated in the neonatal period (between 0 and 28 days of life) within our sector.
* Parents followed in the congenital heart disease sector of the University Hospital of Bordeaux as soon as the diagnosis is announced in antenatal.
* Free, informed and signed written consent of the couple or single mother in a single parent setting or by a third person (in case of physical disability of the participant) and the investigator (no later than the day of inclusion and before any examination required by the research).
* Person affiliated or beneficiary of a social security scheme (excluding AME).
* Parents with parental authority.

Exclusion Criteria:

* Parents who do not understand or read French and cannot be accompanied by a third party for translation.
* Parents with major psychiatric disorders.
* Parents deprived of liberty due to ongoing legal proceedings.
* Parents under guardianship or curatorship or unable to personally express consent.

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2027-02-06 (Estimated); Study Completion 2027-02-06 (Estimated)

PRIMARY OUTCOMES:
Families participation evaluation | at the last protocol visit ( visit 6 - day 180)
  The participation of families in the proposed accompaniment will be evaluated by the participation rate: number of parents who participated in the study until the last stage of the protocol, number of parents who dropped out of the study and reason.

SECONDARY OUTCOMES:
Parental stress Evolution | between visit 1 (day -28) and visit 6 (day 180)
  Evolution of parental stress by the ISP-4 self-questionnaire (Parental Stress Index)
Infant development | at the last protocol visit ( visit 6 - day 180)
  Evolution of the overall score of the Bayley-4 scale (Bayley Infant and Young Child Development Scales) at 6 months of life compared to a literature cohort (neonate child).
Evaluation of the healthcare team adherence | at visit 5 ( day 60 )
  Evaluation of the adherence of the healthcare team to this new model via a Likert scale administered at the discharge of the child, and an analysis of the large items found on the accompanying sheets
Evaluation of the healthcare team adherence | at visit 5 ( day 60 )
  Evaluation of the adherence of the healthcare team to this new model via an EVA scale administered at the discharge of the child, and an analysis of the large items found on the accompanying sheets
Personal Support Project Evaluation | at the last protocol visit ( visit 6 - day 180)
  Evaluation of the Personal Support Project by families using an Visual Analogue Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Cardiologique Haut-Lévêque, Pessac, France, France